CLINICAL TRIAL: NCT01744093
Title: Doxycycline for COPD in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1208012780; R34HL117352 (NIH)
Record Dates: First submitted 2012-11-20; First posted 2012-12-06 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: HIV; Chronic Obstructive Pulmonary Disease (COPD); Emphysema
Keywords: HIV; COPD; Chronic Obstructive Pulmonary Disease; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Doxycycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Doxycycline (Active Comparator): 100 mg twice daily (BID orally) x 24 weeks
  Interventions: Drug: Doxycycline
- Placebo (sugar pill) (Placebo Comparator): 100 mg twice daily (BID orally) x 24 weeks
  Interventions: Drug: Placebo (sugar pill)

INTERVENTIONS:
Drug: Doxycycline — 100 mg twice daily (BID orally) x 24 weeks
  Other Names: Vibramycin
  Arms: Doxycycline
Drug: Placebo (sugar pill) — 100 mg twice daily (BID orally) x 24 weeks
  Other Names: Placebo
  Arms: Placebo (sugar pill)

SUMMARY:
In the context of improved survival from HIV infection itself, chronic obstructive pulmonary disease (COPD); a form of lung disease that includes emphysema, which makes breathing difficult) is emerging as an important cause of morbidity and perhaps ultimately mortality in this population. HIV-infected patients are at increased risk of chronic obstructive pulmonary disease, likely due to multiple factors, including an increased presence of smoking, chronic inflammation and progression of immunodeficiency, oxidant stress (excessive levels of natural chemicals called oxidants and free radicals that can damage tissue), and respiratory infections. While natural history data on COPD are limited in the era of potent antiretroviral therapy, earlier data suggest that the course of emphysema may be accelerated in this population. Our preliminary data suggest that several matrix metalloproteinases (MMPs) derived from alveolar macrophages (a type of immune cell found in the lungs) have an increased cellular response in HIV-infected smokers, which could contribute to accelerated emphysema. Matrix metalloproteinases are enzymes that break down the structural support of tissues, including the airways in the lung.

Based on these observations, the investigators hypothesize that pharmacologic inhibition of matrix metalloproteinases by doxycycline will favorably modify the natural history of chronic obstructive pulmonary disease in HIV-infected patients. To test this hypothesis, the investigators propose conducting a proof of concept pilot study as a prelude to a possible phase II randomized, placebo-controlled trial (testing safety and efficacy in a larger population controlled with a "sugar pill") of doxycycline for COPD in HIV-infected patients should the proof of concept be successful. Our research team is lead by a pulmonologist/researcher with expertise in HIV-associated COPD and an infectious diseases specialist/clinical trials expert.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is emerging as an important cause of morbidity in HIV-infected patients, likely due to multiple factors, including an increased prevalence of smoking, chronic inflammation and immune activation, oxidant stress and respiratory infections. Our preliminary data suggest that several lung matrix metalloproteinases (MMPs) are upregulated in HIV-infected smokers, which could contribute to accelerated emphysema by virtue of their ability to degrade extracellular matrix and basement membrane components. Our Specific Aim is to determine the safety, tolerability, and biologic effects of twice daily doxycycline for 6 months in HIV-infected subjects with COPD. To address this aim, we will conduct a randomized, double-blind, placebo-controlled pilot study of doxycycline 100 mg twice daily in 30 HIV-infected subjects with COPD (2:1 doxy:placebo). The primary endpoint will be safety/tolerability and secondary endpoints will include change in FEV1, reduction of MMP activity in epithelial lining fluid and cells obtained by bronchoscopy and doxycycline levels in blood, ELF and bronchoalveolar lavage (BAL) cell pellets. In addition to providing novel insights into the biologic effects of doxycycline in the lung, the pilot study will inform selection of endpoints for a phase II trial, which ultimately will address an unmet medical need for novel interventions for COPD/emphysema in HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV infection
2. CD4 cell count greater than 200 cells/mm3
3. HIV RNA less than 400 copies/ml
4. Stable antiretroviral therapy for greater than or equal to 12 weeks
5. Fulfills GOLD definition for COPD (post-bronchodilator FEV1/FVC less than 0.7) and/or has radiographic evidence of emphysema
6. Current or history of smoking with minimum 3 pack-year history
7. ALT and AST less than 3 x upper limit of normal
8. For women of childbearing potential: willingness to use 2 forms of birth control
9. Subjects on therapy for COPD must be on stable therapy for at least 4 weeks

Exclusion Criteria:

1. Pulmonary infection, COPD exacerbation, or acute opportunistic infection within 30 days of entry
2. Conditions associated with increased sedation of bronchoscopy risk, including but not limited to Gold class 3 or 4 COPD, requirement for home oxygen, hypercapneic respiratory failure, poorly controlled hypertension
3. Known allergy/intolerance to doxycycline, atropine, or any local anesthetic
4. Inability to provide informed consent
5. Pregnant or lactating women
6. Men must agree not to attempt to make a woman pregnant or participate in sperm donation during the study and for 6 weeks after discontinuing the drug
7. End stage renal disease
8. Cirrhosis
9. INR greater than 1.4
10. Platelets less than 80,000
11. Any condition including active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or increase the risk of bronchoscopy
12. Active or planned participation in any other clinical trial or observational study without prior approval from the PI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kaner, MD, Principal Investigator — Weill Cornell Medical College-New York Presbyterian Hospital; Marshall Glesby, MD, Principal Investigator — Weill Cornell Medical College-New York Presbyterian Hospital
Locations (1):
- Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 61 subjects enrolled into the study, 34 subjects did not pass screening.
Groups:
- Doxycycline: Doxycycline x 100 mg twice daily (BID orally) for 24 weeks
- Placebo (Sugar Pill): One pill twice daily (BID orally) for 24 weeks
Period: Overall Study
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Started | 18 | 9
Treated | 16 | 8
Completed | 12 | 8
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Doxycycline: Doxycycline x 100 mg BID (orally) for 24 weeks
- Placebo (Sugar Pill): Placebo (sugar pill) x 100 mg BID (orally) for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 9 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 16 | 9 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 4 | 2 | 6
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety of Doxycycline, as Measured by the Number of Subjects With Any Treatment-related Adverse Events.
Description: To determine the safety of twice daily doxycycline for 24 weeks in HIV-infected subjects with COPD and/or emphysema as measured by the number of subjects with any treatment-related adverse events.
Time Frame: Up to 24 weeks
Population: 2 subjects were randomized to the doxycycline arm, but withdrew prior to starting the study drug. 1 subject was randomized to the placebo arm, but withdrew prior to starting the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 16 | 8
Participants | 3 | 1
Statistical Analysis 1: Comparison: Doxycycline; Test type: Other — Descriptive proportion; Proportion (percent) = 18.8, 95% CI 2-sided [4.0 to 45.6] — Exact two-sided 95% Clopper-Pearson confidence interval

2. Primary Outcome: Tolerability of Doxycycline, as Measured by the Number of Subjects With a Dose-limiting Toxicity
Description: To determine the tolerability of twice daily doxycycline for 24 weeks in HIV-infected subjects with COPD and/or emphysema as measured by those subjects experiencing a dose-limiting toxicity
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 16 | 8
Participants | 1 | 1
Statistical Analysis 1: Comparison: Doxycycline; Null hypothesis adverse event rate (grade 2 or higher toxicity) = 45.5%; Test type: Superiority; p = 0.002, Fisher Exact; Proportion (percent) = 6.3, 95% CI 2-sided [0.16 to 30.2] — Exact two-sided 95% Clopper-Pearson confidence interval

3. Secondary Outcome: Clinical: Change in Pulmonary Function (FEV1)
Description: FEV1 is the volume of air exhaled during the first second of a forced expiratory maneuver.
Time Frame: 24 Weeks
Population: At 24 Weeks, total 7 subjects were not analyzed at Week 24. With arm-Doxycycline, 6 subjects dropped out; with arm-Placebo, 1 subject dropped out.
Measure: Median (Inter-Quartile Range); unit: Percentage of predicted FEV1
Groups:
- Placebo (Sugar Pill): One pill twice daily (BID orally) x 24 Weeks
  Placebo (sugar pill): One pill twice daily (BID orally) x 24 Weeks
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 12 | 8
Percentage of predicted FEV1 | -1.5 [-4.5 to 2.25] | 1 [-1.75 to 5]

4. Secondary Outcome: Percent Change in BAL MMP-9 Activity
Description: Percent change of MMP-9 activity in bronchoalveolar lavage (BAL) fluid.
Time Frame: 12 Weeks
Population: With arm-Doxy, 8 subjects were not analyzed at Week 12 because 5 subjects dropped out, 2 subjects had an inadequate sample, 1 subject could not have the bronchoscopy. With arm-Placebo, 2 subjects were not analyzed at Week 12 because 1 subject dropped out and 1 subject could not have the bronchoscopy.
Measure: Median (Inter-Quartile Range); unit: Percent change
Groups:
- Placebo (Sugar Pill): One pill twice daily (BID orally) x 24 Weeks
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 10 | 7
Percent change | -42 [-62 to -28] | 21 [-23 to 93]

5. Secondary Outcome: Doxycycline Levels
Description: Doxycycline level in serum
Time Frame: 12 Weeks
Population: With arm-Doxy, 6 subjects were not analyzed at Week 12 because 5 subjects dropped out, 1 subject did not provide a sample. With arm-Placebo, 2 subjects were not analyzed at Week 12 because 1 subject dropped out and 1 subject did not provide a sample.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Placebo (Sugar Pill): One pill (BID orally) x 24 Weeks
  Placebo (sugar pill): One pill twice daily (BID orally) x 24 Weeks
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 12 | 7
ng/ml | 3005 [2684 to 4179] | 0 [0 to 0]

6. Secondary Outcome: Doxycycline Levels in BAL
Description: Doxycycline levels in bronchoalveolar lavage (BAL) fluid.
Time Frame: 12 Week
Population: With arm-Doxy, 6 subjects were not analyzed at Week 12 because 5 subjects dropped out, 1 subject could not have the bronchoscopy. With arm-Placebo, 2 subjects were not analyzed at Week 12 because 1 subject dropped out and 1 subject could not have the bronchoscopy.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Doxycycline | Placebo (Sugar Pill)
Number analyzed (Participants) | 12 | 7
ng/ml | 16.75 [10.88 to 22.15] | 0 [00 to 00]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Clinical assessments included full physical examination at screening, targeted physical examinations at other visits, ongoing assessments for adverse events and new clinical diagnoses and CAT review at each visit. Safety labs were obtained at weeks 2, 6, 12, 18, and 24. 2 participants in the doxycycline arm and 1 participant in the placebo arm were not evaluated for adverse events because they did not take the study drug.
Arm/Group | Doxycycline | Placebo (Sugar Pill)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 13/16 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=16) | Placebo (Sugar Pill) (N=8)
Oral thrush (Infections and infestations) | 1 (1) | 0 (0)
Hemoglobin drop (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mouth lesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Excoriated lesions on arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Intermittent diarrhea for 4-5 wk (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scattered maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemoptysis (mild) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Low absolute neutrophil count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain on right side (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT01744093/Prot_SAP_000.pdf